CLINICAL TRIAL: NCT05657392
Title: Examination of Changes in Quantitative EEG Parameters Based on Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment in Patients With Post Stroke
Brief Title: Quantitative EEG Changes Following Repetitive Transcranial Magnetic Stimulation in Patients With Post Stroke (EEG-rTMS)
Acronym: EEG-rTMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Onan Güren, Asst. Prof. Dr., Izmir Katip Celebi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-KAE-0017; 120E512 (Other Grant/Funding Number: THE SCIENTIFIC AND TECHNOLOGICAL RESEARCH COUNCIL OF TURKEY); 2022-TDR-MÜMF-0014 (Other Grant/Funding Number: IKCU Scientific Research Projects Coordination Unit); 2021-ÖDL-MÜMF-0004 (Other Grant/Funding Number: IKCU Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2022-11-26; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Stroke; Stroke, Ischemic; Stroke/Brain Attack
Keywords: Post Stroke; Repetitive Transcranial Magnetic Stimulation; Motor Recovery; quantitative EEG; Electroencephalogram; biomarkers
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inhibitory repetitive Transcranial Magnetic Stimulation (Experimental): All patients will receive inhibitory repetitive transcranial magnetic stimulation (rTMS) treatment at 1 Hz frequency. The contralesional primary motor cortex region will be stimulated with a Neurosoft-Neuro MS/D device. There will be a total of 10 treatment sessions over a 2-week period. Before each intervention, the resting motor threshold (rMT) value will be determined. rMT will be detected by obtaining a motor-evoked potential of >50 μV amplitude on EMG recording of the contralateral first dorsal interosseous muscle in at least 5 out of 10 stimulations to the primary motor cortex. 90% of the motor threshold will be set in the stimulation. Each stimulation is planned for a total of 20 minutes and a total of 1200 pulses in the form of 1 Hz stimulation.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS); Other: 32 electrode electroencephalography (EEG)

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation (rTMS) — Repetitive Transcranial Magnetic Stimulation (rTMS) is a noninvasive intervention that uses magnetic fields to stimulate nerve cells to improve the symptoms of a variety of disorders, including stroke-related motor impairment. Last few decades, it has been revealed that rTMS accelerates motor recovery and may reduce stroke-related symptoms.
Other: 32 electrode electroencephalography (EEG) — 32-electrode EEG will be non-invasively recorded from electrodes placed in a montage over the scalp while the participant is resting

SUMMARY:
Quantitative EEG (qEEG) has been used as an effective tool in the diagnosis and prognosis of brain-related diseases. In the literature, a variety of qEEG parameters have been proven informative in the prognosis of stroke. In addition, it has been demonstrated that changes in certain qEEG parameters during traditional/task-specific rehabilitation approaches are correlated with clinical outcomes of functional motor recovery. Repetitive transcranial magnetic stimulation (rTMS) has been proposed as a non-invasive and therapeutic treatment used to accelerate and enhance the recovery process of motor function in stroke patients. Many studies have reported that inhibiting contralesional rTMS may have positive effects in stroke patients with severe upper extremity motor impairment. In this context, the aim of the proposed study is to investigate whether there is a correlation between the change in qEEG parameters and the improvement of motor functions associated with rTMS treatment and to provide an electrophysiological prognostic biomarker of inhibiting contralesional rTMS for stroke patients.

DETAILED DESCRIPTION:
50 stroke patients will receive inhibiting contralesional rTMS at 1 Hz frequency. Upper extremity motor functions will be assessed with Fugl-Meyer Assessment-Upper Extremities (FMA-UE), Brunnstrom stages, modified Ashworth Scale (MAS) before and after treatment. The resting-state EEGs will be measured six time during the course of the treatment (Before/After 1. Session, Before/After 5. Session, Before/After 10. Session (end of the treatment)).

The main questions it aims to answer are:

50 stroke patients will receive inhibiting contralesional rTMS at 1 Hz frequency. Upper extremity motor functions will be assessed with Fugl-Meyer Assessment-Upper Extremities (FMA-UE), Brunnstrom stages, modified Ashworth Scale (MAS) before and after treatment. The resting-state EEGs will be measured six time during the course of the treatment (Before/After 1. Session, Before/After 5. Session, Before/After 10. Session (end of the treatment)).

The main questions it aims to answer are:

1. How do the previously suggested quantitative EEG parameters (decrease in DAR (Delta Alpha power ratio), BSI (Brain Symmetry Index) and DTAB (Delta-theta to alpha-beta ratio, increase in alpha mean frequency ) change with rTMS application for the recovery of motor functions in patients with stroke and can they be defined as an effective biomarker for stroke treatment with rTMS?
2. Can the clinical response to rTMS be estimated from the quantitative EEG parameters calculated from just before rTMS application?
3. Can electrophysiological effect of rTMS be observed from EEG measurements throughout the application?

ELIGIBILITY:
Inclusion Criteria:

* Older than age of 18 years.
* Presence of ischemic or hemorrhagic stroke confirmed by MRI.
* Having a stroke for the first time.
* Patients who agreed to participate by signing the informed consent form.

Exclusion Criteria:

* Presence of a clinical condition (metallic implant, cardiac or brain pace, claustrophobia, head trauma, cranial operation history) that may constitute a contraindication to repetitive transcranial magnetic stimulation intervention.
* Presence of malignancy or systemic rheumatic disease
* Pregnancy or breastfeeding
* Non-stroke disease or lesion affecting the sensorimotor system
* Alcohol or drug addiction
* Presence of pump/shunt
* Presence of severe cognitive impairment
* Presence of >3 spasticity in the upper extremity defined according to the Modified Ashworth Scale
* History of psychiatric illness such as major depression/personality disorders
* History of epilepsy or taking medication due to epilepsy
* Diagnosed with dementia
* Received rTMS intervention before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in The Fugl-Meyer Assessment (FMA) | (1) Baseline, (2) At the end of the last session of the intervention (immediately after the 10th session, each session is 1 day)
  The Fugl-Meyer Assessment (FMA) is a clinical stroke-specific scale that an assesment sensorimotor impairment. It is a powerful index applied clinically and also in research to identify the stroke severity, determine the motor recovery and to plan the rTMS interventions.

SECONDARY OUTCOMES:
Change in Modified Ashworth Scale | (1) Baseline, (2) At the end of the last session of the intervention (immediately after the 10th session, each session is 1 day)
  The modified Ashworth Scale is a clinical index that used for assessment of muscle tone and evaluates the resistance occuring during passive range of motion.
Change in Brunnstrom Stages of Stroke Recovery | (1) Baseline, (2) At the end of the last session of the intervention (immediately after the 10th session, each session is 1 day)
  The Brunnstrom stages are a clinical scale that describe the changes in the ability of movement and the development and reorganization of brain at the post-stroke stage.

CONTACTS AND LOCATIONS:
Overall Officials: Onan Guren, PhD, Principal Investigator — Izmir Katip Celebi University; Ayhan Askin, MD, Study Director — Izmir Katip Celebi University; Ilker Sengul, MD, Principal Investigator — Izmir Katip Celebi University; Mehmet Akif Ozdemir, PhD Cand., Principal Investigator — Izmir Katip Celebi University
Locations (1):
- Izmir Katip Celebi University, Izmir, Cigli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication All individual (confidential) data including clinical outcomes, demographic and clinical surveys, EEG measurements, MRI data, etc.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: All IPD will be shared with a dataset article.
Access Criteria: Will be announced.

REFERENCES:
- [Background] Alekseichuk I, Mantell K, Shirinpour S, Opitz A. Comparative modeling of transcranial magnetic and electric stimulation in mouse, monkey, and human. Neuroimage. 2019 Jul 1;194:136-148. doi: 10.1016/j.neuroimage.2019.03.044. Epub 2019 Mar 22. PMID 30910725
- [Background] Bembenek JP, Kurczych K, Karli Nski M, Czlonkowska A. The prognostic value of motor-evoked potentials in motor recovery and functional outcome after stroke - a systematic review of the literature. Funct Neurol. 2012 Apr-Jun;27(2):79-84. PMID 23158578
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Byblow WD, Stinear CM, Barber PA, Petoe MA, Ackerley SJ. Proportional recovery after stroke depends on corticomotor integrity. Ann Neurol. 2015 Dec;78(6):848-59. doi: 10.1002/ana.24472. Epub 2015 Nov 17. PMID 26150318
- [Background] Claflin ES, Krishnan C, Khot SP. Emerging treatments for motor rehabilitation after stroke. Neurohospitalist. 2015 Apr;5(2):77-88. doi: 10.1177/1941874414561023. PMID 25829989
- [Background] Conforto AB, Anjos SM, Saposnik G, Mello EA, Nagaya EM, Santos W Jr, Ferreiro KN, Melo ES, Reis FI, Scaff M, Cohen LG. Transcranial magnetic stimulation in mild to severe hemiparesis early after stroke: a proof of principle and novel approach to improve motor function. J Neurol. 2012 Jul;259(7):1399-405. doi: 10.1007/s00415-011-6364-7. Epub 2011 Dec 16. PMID 22173953
- [Background] Coupar F, Pollock A, Rowe P, Weir C, Langhorne P. Predictors of upper limb recovery after stroke: a systematic review and meta-analysis. Clin Rehabil. 2012 Apr;26(4):291-313. doi: 10.1177/0269215511420305. Epub 2011 Oct 24. PMID 22023891
- [Background] Finnigan SP, Rose SE, Walsh M, Griffin M, Janke AL, McMahon KL, Gillies R, Strudwick MW, Pettigrew CM, Semple J, Brown J, Brown P, Chalk JB. Correlation of quantitative EEG in acute ischemic stroke with 30-day NIHSS score: comparison with diffusion and perfusion MRI. Stroke. 2004 Apr;35(4):899-903. doi: 10.1161/01.STR.0000122622.73916.d2. Epub 2004 Mar 4. PMID 15001786
- [Background] Finnigan S, Wong A, Read S. Defining abnormal slow EEG activity in acute ischaemic stroke: Delta/alpha ratio as an optimal QEEG index. Clin Neurophysiol. 2016 Feb;127(2):1452-1459. doi: 10.1016/j.clinph.2015.07.014. Epub 2015 Jul 22. PMID 26251106
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Griskova I, Ruksenas O, Dapsys K, Herpertz S, Hoppner J. The effects of 10 Hz repetitive transcranial magnetic stimulation on resting EEG power spectrum in healthy subjects. Neurosci Lett. 2007 May 29;419(2):162-7. doi: 10.1016/j.neulet.2007.04.030. Epub 2007 Apr 18. PMID 17478041
- [Background] Kobayashi M, Pascual-Leone A. Transcranial magnetic stimulation in neurology. Lancet Neurol. 2003 Mar;2(3):145-56. doi: 10.1016/s1474-4422(03)00321-1. PMID 12849236
- [Background] Langhorne P, Coupar F, Pollock A. Motor recovery after stroke: a systematic review. Lancet Neurol. 2009 Aug;8(8):741-54. doi: 10.1016/S1474-4422(09)70150-4. PMID 19608100
- [Background] Nowak DA, Grefkes C, Ameli M, Fink GR. Interhemispheric competition after stroke: brain stimulation to enhance recovery of function of the affected hand. Neurorehabil Neural Repair. 2009 Sep;23(7):641-56. doi: 10.1177/1545968309336661. Epub 2009 Jun 16. PMID 19531606
- [Background] Wagner T, Valero-Cabre A, Pascual-Leone A. Noninvasive human brain stimulation. Annu Rev Biomed Eng. 2007;9:527-65. doi: 10.1146/annurev.bioeng.9.061206.133100. PMID 17444810